CLINICAL TRIAL: NCT01744418
Title: A Pilot Study for Evaluation of the Safety and Efficacy of Humacyte's Human Acellular Vascular Graft for Use as a Vascular Prosthesis for Hemodialysis Access in Patients With End-Stage Renal Disease
Brief Title: Evaluation of the Safety and Efficacy of a Vascular Prosthesis for Hemodialysis Access in Patients With ESRD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Humacyte, Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN-PRO-V001
Record Dates: First submitted 2012-12-05; First posted 2012-12-06 (Estimated); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: End-stage Renal Disease; Kidney Failure, Chronic
Keywords: ESRD; HEMODIALYSIS; CHRONIC RENAL INSUFFICIENCY; Renal Dialysis; Hemodiafiltration; Blood Vessel Prosthesis; Tissue-Engineered Vascular Graft; Vascular Prosthesis Implantation
MeSH Terms: conditions — Kidney Failure, Chronic; Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HAVG graft (Experimental): HAVG graft implantation to study participants.
  Interventions: Device: HAVG graft implantation

INTERVENTIONS:
Device: HAVG graft implantation — Patients will be implanted with a Human Acellular Vascular Graft (HAVG) in the forearm or upper arm (arterial anastomosis to the radial or brachial artery, venous anastomosis to either the brachial, cephalic or very central basilica vein) using standard vascular surgical techniques. The graft will be placed in a straight or curved configuration in the first 10 patients. Loop grafts may be permitted in subsequent patients subject to acceptable graft performance at the interim safety review. Placing the graft across the elbow will be avoided.
  Other Names: Human Acellular Vascular Graft

SUMMARY:
The purpose of this study is to assess the safety and efficacy of a novel, tissue-engineered vascular prosthesis, the Human Acellular Vascular Graft, HAVG.

The HAVG is intended as an alternative to synthetic materials and to autologous grafts in the creation of vascular access for dialysis.

DETAILED DESCRIPTION:
The HAVG is a sterile, non-pyrogenic, acellular tubular graft composed of human collagens and other natural extra-cellular matrix proteins. Upon implantation, it is anticipated (based on pre-clinical studies) that the collagen-based matrix comprising the graft will be infiltrated with host cells and re-modeled by the host. This will result in a vascular structure more similar to the histological composition of the native vascular tissue that may improve graft longevity and be less likely to become infected.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end stage renal disease (ESRD) who are not, or who are no longer, candidates for creation of an autogenous AV fistula and therefore need placement of an AV graft in the upper extremity to start or maintain hemodialysis therapy
* Patients between 18 and 75 years old, inclusive
* Suitable anatomy for implantation of straight forearm grafts or curved upper arm grafts (arterial anastomosis to radial or brachial artery, venous anastomosis to either brachial cephalic or very central basilica vein)
* Hemoglobin ≥8g/dL and platelet count ≥100,000/mm3 prior to Day 1
* Other hematological and biochemical parameters within a range consistent with ESRD and acceptable for the administration of general anesthesia prior to Day 1
* Adequate liver function, defined as serum bilirubin ≤1.5 mg/dL; GGT, AST, ALT, and alkaline phosphatase ≤2x upper limit of normal or INR ≤ 1.5 prior to Day 1.
* Ability to communicate meaningfully with investigative staff, competence to give written informed consent, and ability to comply with entire study procedures
* Able and willing to give informed consent
* Life expectancy of at least 1 year

Exclusion Criteria:

* History or evidence of severe cardiac disease (NYHA Functional Class III or IV), myocardial infarction within six months of study entry (Day 1), ventricular tachyarrhythmias requiring continuing treatment, or unstable angina
* History or evidence of severe peripheral vascular disease in the upper limbs
* Known or suspected central vein obstruction on the side of planned graft implantation
* Stroke within six (6) months of study entry (Day 1)
* Treatment with any investigational drug or device within 60 days prior to study entry (Day 1)
* Treatment with vitamin K-antagonists or direct thrombin inhibitors within the previous month to study entry (Day 1)
* All patients (including both female patients of childbearing potential and male patients with childbearing potential partners) who do not use a highly effective method of birth control (failure rate less than 1% per year when used consistently and correctly), e.g. implants, injectables, combined oral contraceptives in combination with a barrier method, some intrauterine contraceptive devices, sexual abstinence, or a vasectomized partner
* Active diagnosis of cancer within the previous year
* Immunodeficiency including AIDS / HIV
* Documented hypercoagulable state or history of 2 or more DVTs or other spontaneous intravascular thrombotic events
* Bleeding diathesis
* Active autoimmune disease
* Previous PTFE graft in the operative limb unless the HAVG can be placed more proximally than the previous failed graft
* More than 1 failed PTFE graft in the operative limb
* Active local or systemic infection (WBC > 15,000/mm3)
* Patients receiving a forearm graft with which crosses the elbow
* Patients receiving an upper arm graft with arterial anastomosis to the axillary artery or venous anastomosis to the axillary vein
* Patients receiving a lower extremity AV access
* Known serious allergy to aspirin or penicillin
* Any other condition which in the judgment of the investigator would preclude adequate evaluation of the safety and efficacy of the HAVG
* Previous enrollment in this study
* Employees of the sponsor or patients who are employees or relatives of the investigator
* PRA > 20% (first 10 patients only)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-11-22 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
HAVG safety & tolerability | At each visit within first 6 months after HAVG implantation.
  The incidence of aneurysm formation, anastomotic bleeding or rupture, graft infection and irritation/inflammation/infection at the implantation site will be tabulated by visit and overall.
HAVG patency rate | At 6 months after HAVG implantation.
  Determine the patency (primary, primary assisted and secondary) rate of the Humacyte HAVG.

SECONDARY OUTCOMES:
PRA response | At screening, day 15, 29, 57 and week 12, 26
  Assess changes in the PRA response over the 6 months after graft implantation.
IgG antibodies | At screening, day 15, 29, 57 and week 12, 26
  Determine whether IgG antibodies to the extracellular matrix material are formed in response to implantation of the HAVG.
Patency maintenance/restoration | At each visit except screening.
  Determine the rates of interventions needed to maintain / restore patency in the graft.
HAVG patency rates | At 12, 18, 24 months after HAVG implantation.
  Patency rates (primary, primary assisted and secondary) at 12, 18 and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Shamik Parikh, MD, Study Director — Humacyte, Inc.
Locations (3):
- Poland (3):
  - Department of Vascular Surgery and Angiology at the Medical University Lublin, Lublin
  - Independent Public Central Clinical Hospital in Warsaw; Department of General, Vascular and Transplant Surgery, Warsaw
  - Regional Specialist Hospital in Wroclaw; Clinic of Vascular Surgery, Wroclaw

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lawson JH, Glickman MH, Ilzecki M, Jakimowicz T, Jaroszynski A, Peden EK, Pilgrim AJ, Prichard HL, Guziewicz M, Przywara S, Szmidt J, Turek J, Witkiewicz W, Zapotoczny N, Zubilewicz T, Niklason LE. Bioengineered human acellular vessels for dialysis access in patients with end-stage renal disease: two phase 2 single-arm trials. Lancet. 2016 May 14;387(10032):2026-34. doi: 10.1016/S0140-6736(16)00557-2. PMID 27203778
- See also: Results of the clinical study have been published — https://pubmed.ncbi.nlm.nih.gov/27203778/